CLINICAL TRIAL: NCT05170698
Title: Coalition Excision and Corrective Osteotomies vs Coalition Excision and Arthroereisis in Management of Pes Planovalgus With Talocalcaneal Coalition in Adolescent
Brief Title: Management of Pes Planovalgus With Talocalcaneal Coalition ,Osteotomy vs Arthroereisis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 0000017585
Record Dates: First submitted 2021-06-27; First posted 2021-12-28 (Actual); Last update posted 2022-06-03 (Actual); Status verified 2022-06

CONDITIONS: Talocalcaneal Bar; Pes Planus
MeSH Terms: conditions — Flatfoot

STUDY DESIGN:
Intervention Model Description: 2 groups one with the first intervention arthroereisis and bar excision the second with bar excision and osteotomies it may be one or multiple
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- coalition excision and arthroereisis (Experimental): Talocalcaneal bar excision is done and then arthroereisis implant is applied in subtalar joint to correct rigid pes planovalgus in adolescent
  Interventions: Procedure: Coaltion excision and arthroereisis
- coalition excision and corrective osteotomies (Experimental): Talocalcaneal bar excision is done and then according to degree of deformity either medial displacement calcaneal osteotomy or evans or cotton osteotomy is done or combined together to correct rigid pes planovalgus in adolescents
  Interventions: Procedure: Coalition excision and corrective osteotomies

INTERVENTIONS:
Procedure: Coaltion excision and arthroereisis — Both done to treat rigid flat foot with talocalcaneal coalition. Talocalcaneal coalition excision and management of rigid pes planovalgus in adolescent
  Other Names: Coalition excision and corrective osteotomies
  Arms: coalition excision and arthroereisis
Procedure: Coalition excision and corrective osteotomies — Both done to treat rigid flat foot with talocalcaneal coalition. Talocalcaneal coalition excision and management of rigid pes planovalgus in adolescent
  Arms: coalition excision and corrective osteotomies

SUMMARY:
the investigators compare the corrective osteotomies vs arthroereisis in management of talcalcaneal coalition in adolescents as regard the outcome to provide the best intervention for the patient

DETAILED DESCRIPTION:
In talocalcaneal coalition management is controversial so in this study the invstigators try to compare techniques other than coalition excision only or fusion only by using two types of intervention including first coalition excision and multiple corrective osteotomies according to deformity as evans ,medial displacement calcaneal osteotomy and cotton osteotomy vs coalition excision and arthroereisis the investigators compare functional and radiological outcomes and complication to provide the best management for these patients .

ELIGIBILITY:
Inclusion Criteria:

* flat foot due to talocalcaneal coalition Symptomatic patient Resectable coalition Age between 10 and 20

Exclusion Criteria:

* flat foot of other etiology Age more than 20 Concurrent knee deformity unless corrected before surgery Extensive coalition more than 50 %of posterior facet

Ages: 10 Years to 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2018-11-18 (Actual); Primary Completion 2021-12-18 (Actual); Study Completion 2021-12-30 (Actual)

PRIMARY OUTCOMES:
Degree of deformity valgus | preoperative
  By goniometer
Degree of deformity valgus | three months
  By goniometer
Degree of deformity valgus | six months
  By goniometer
Degree of deformity valgus | one year postoperative
  By goniometer
Degree of deformity valgus | two year postoperative
  By goniometer
Subtalar range of motion | preoperative
  By geniometer for inversion and eversion
Subtalar range of motion | three months
  By geniometer for inversion and eversion
Subtalar range of motion | six months
  By geniometer for inversion and eversion
Subtalar range of motion | one year postoperative
  By geniometer for inversion and eversion
Subtalar range of motion | two year postoperative
  By geniometer for inversion and eversion

SECONDARY OUTCOMES:
functional outcome | preoperative
  By foot ankle ability measurement score
Patient satisfaction | preoperative
  By foot and ankle disability score
functional outcome | three months
  By foot ankle ability measurement score
Patient satisfaction | three months
  By foot and ankle disability score
functional outcome | six months
  By foot ankle ability measurement score
Patient satisfaction | six months
  By foot and ankle disability score
functional outcome | one year
  By foot ankle ability measurement score
functional outcome | two year
  By foot ankle ability measurement score
Patient satisfaction | one year
  By foot and ankle disability score
Patient satisfaction | two year
  By foot and ankle disability score

OTHER OUTCOMES:
AOFAS | preoperative
  he American Orthopaedic Foot & Ankle Society (AOFAS) score up to 100 the higher the score the better function
AOFAS | three months
  he American Orthopaedic Foot & Ankle Society (AOFAS) score up to 100 the higher the score the better function
AOFAS | six months
  he American Orthopaedic Foot & Ankle Society (AOFAS) score up to 100 the higher the score the better function
AOFAS | one year
  he American Orthopaedic Foot & Ankle Society (AOFAS) score up to 100 the higher the score the better function
AOFAS | two year
  he American Orthopaedic Foot & Ankle Society (AOFAS) score up to 100 the higher the score the better function

CONTACTS AND LOCATIONS:
Overall Officials: ayman m howeidy, professor, Study Chair — Ain Shams University
Locations (1):
- Ain shams university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] El Shazly O, Mokhtar M, Abdelatif N, Hegazy M, El Hilaly R, El Zohairy A, Tawfik E. Coalition resection and medial displacement calcaneal osteotomy for treatment of symptomatic talocalcaneal coalition: functional and clinical outcome. Int Orthop. 2014 Dec;38(12):2513-7. doi: 10.1007/s00264-014-2535-3. Epub 2014 Sep 25. PMID 25248861
- [Background] Siddiqui NA, Lamm BM. Digital planning for foot and ankle deformity correction: Evans osteotomy. J Foot Ankle Surg. 2014 Nov-Dec;53(6):700-5. doi: 10.1053/j.jfas.2014.04.011. Epub 2014 Jun 6. PMID 24909804